# **Document Coversheet**

Study Title: Randomized Trial of a Social Media-Delivered Intervention

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 8/29/2024 |
| NCT Number: | NCT03441321 |
| IRB Number | 56153 |
| Coversheet created: | 2/4/2025 |

## Survey Cover Letter Consent

Researchers at the University of Kentucky are inviting you to take part in an online study. In the study, participants complete online surveys and join a Facebook group which posts information to start conversations that promote physical and mental wellness and healthy lifestyles. The goal of the study is to understand participants' views of the group and conversation topics.

The information provided on this screen will help you decide whether you want to take part in this study. It is your choice to take part or not.

WHAT IS MY INVOLVEMENT IN THIS STUDY AND HOW LONG WILL IT LAST? There are several steps in this study:

- 1. After you finish reading this study information page, you will complete an initial online survey that will take about 30 minutes and asks questions about your use of social media, your health behaviors, and your thoughts about your life style habits.
- 2. You will then be invited to join one of two private and hidden Facebook groups with similar content. Once the Facebook group is established, the moderator will begin to regularly post content twice a day for 8 weeks. Each week will focus on a different theme. We ask that you check the Facebook group each day, read the content, provide reactions (for example, clicking "like"), add your comments to discussions within the secret group, and share you own relatedposts.
- 3. Complete additional online surveys after the group concludes. These surveys will be emailed to you 3, 8 and 18 months after completing the first survey. These surveys will take approximately 30 minutes to complete and will contain similar questions to the first survey as well as some questions that ask for your opinions of the Facebook group experience.

#### WILL I GET PAID TO PARTICIPATE?

Yes. We will email you the redemption code for a \$30 Amazon gift card after you finish the initial survey and additional \$30 gift cards after the completion of each of the 3 and 8-month surveys. You will receive a \$40 gift card for completing the 18-month survey. We will not provide any compensation for participating in the Facebook group. You could be paid a total of \$130 for completing all parts of the study.

#### ARE THERE ANY BENEFITS TO ME IF I CHOOSE TO TAKE PART IN THIS STUDY?

There may be no direct benefit to you from participating in this research. However, your responses may help us understand more about how to improve educational and prevention programs designed to promote healthy lifestyles. Some volunteers experience satisfaction from knowing they have contributed to research that may possibly benefit others in the future.

#### WHAT ARE THE RISKS OR DISCOMFORTS I MIGHT EXPERIENCE IF I TAKE PART IN THIS STUDY?

The potential risks of this study are minimal. Some questions may make you upset or feel uncomfortable, although we have attempted to minimize this, and you may choose not to answer or respond to them. If some questions do upset you, we can tell you about some people who may be able to help you with these feelings. You are also free to quit the research study at any time.

#### HOW WILL MY INFORMATION BE KEPT PRIVATE OR CONFIDENTIAL?

Your response to the survey will be kept confidential to the extent allowed by law. When we write about the study you will not be identified.

Please be aware, while we make every effort to safeguard your data once received on our servers via Qualtrics, given the nature of online surveys, as with anything involving the Internet, we can never guarantee the confidentiality of the data while still en route to us. We will not ask you to provide your name on the survey data collection in order to keep your identity separate from your research data. Your identifiable information collected at the start of the study will not be stored with your responses. Instead, your responses will be assigned a subject number which will be stored separately from your responses so others will not know which responses are yours. We will securely store the key code linking your responses to your identifiable information in a separate password protected file which will be destroyed two years after the study is completed.

You will be invited to join a private and hidden Facebook group where only other members participating in the study and study researchers will have access. Your responses to postings in the group are visible only to group members. Study researchers and other group members will not have access to your personal Facebook profile or any information beyond that which you have made publicly available on your personal profile (unless you "friend" other participants which is not required for participation). Any postings that you make in the group will be visible to other members so please do not post any personal or health related information that you are uncomfortable with sharing. We will use data from your interactions within the Facebook group including when you view, like, or comment on a post. We will not obtain data from your personalprofile or posts you make outside of the group.

We will download data from the private and hidden Facebook group including posts, comments, and reactions from the moderator, you, and other people in the group so that we can study this data to better understand how people participated. We will not download any data from your Facebook profile. The research team will not download any photographs you share in the Facebookgroup when we download engagement data. Facebook may ask you to indicate (for example, by clicking on a button) that you are OK with us collecting these data from Facebook.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National

Institutes of Health. The researchers will use this Certificate to legally refuse to disclose any information, documents or biospecimens that may identify you, including from a court order. This means that research material collected about you for this study will not be released to anyone whois not connected with this study unless:

- you request or consent to its release;
- a law requires its release (such as reporting communicable diseases or child abuse to Stateagencies);
- it is used for other scientific research, as allowed by federal regulations protecting subjects; or
- it is requested by the U.S. federal or state agency sponsoring the research that is neededfor auditing or program evaluation or to meet the requirements of the Food and Drug Administration (FDA).

### WHAT WILL HAPPEN TO INFORMATION I PROVIDE IN THE RESEARCH AFTER THE STUDY IS OVER?

Identifiable information such as your name and contact information may be removed from the information collected in this study. After removal of your identifiable information, the information may be used for future research or shared with other researchers without your additional informed consent.

WHAT WILL HAPPEN IF I DO NOT WANT TO TAKE PART OR DECIDE LATER TO NOT STAY IN THE STUDY?

We hope to receive have about 400 people participate in the study, so your answers are important to us. Of course, you have a choice about whether or not to complete this survey/questionnaire as well as any future study activities, but if you do participate, you are free to skip any questions or discontinue at any time.

THE RESEARCH TEAM HAS THE RIGHT TO REMOVE YOU FROM THE STUDY AT ANYTIME.

The University of Kentucky does not tolerate profanity, vulgarity, personal attacks, trolling, discrimination, and any posts that inflame hot topics such as, but not limited to, religion and politics in the Facebook group. In the event we find these posts during the study, we will remove them and give you a warning. If this continues to become an issue in the group, we will remove you from the group and withdraw you from participation and future compensation. You cannot complete the survey more than once or you will not receive compensation and will be removed from the study. We will also remove you from the study if you provide responses to our surveys that fail our quality assurance checks designed to detect bots and fake survey responses.

WHO CAN I CALL IF I HAVE ANY QUESTIONS ABOUT THE STUDY?

If you have questions about the study, please feel free to ask; my contact information is given below. If you

have complaints, suggestions, or questions about your rights as a research volunteer, contact the staff in the University of Kentucky Office of Research Integrity at 859-257-9428 or toll-free at 1-866-400-9428

Thank you in advance for your assistance with this important project.

Sincerely

Jerod Stapleton, Ph.D.

Department of Health, Behavior & Society/College of Public Health, University of Kentucky

PHONE: 859-562-2802

E-MAIL: jerod.stapleton@uky.edu

By beginning this research, I acknowledge that I am 18 years of age or older and have read and understand the information. I agree to take part in the research, with the knowledge that I am free to withdraw my participation in the research without penalty.

Click on the "I Agree" button to confirm your agreement to take part in the research and begin taking the survey.

I Agree I Do Not Agree